CLINICAL TRIAL: NCT04948866
Title: Palliative Care for Persons With Late-stage Alzheimer's and Related Dementias and Their Caregivers
Acronym: ADRD-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-2764; R01AG065394 (NIH)
Record Dates: First submitted 2021-06-23; First posted 2021-07-02 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Dementia, Vascular; Dementia With Lewy Bodies; Dementia Frontal; Dementia, Mixed; Dementia Alzheimers; Alzheimer Disease; Dementia Severe
MeSH Terms: conditions — Dementia; Dementia, Vascular; Lewy Body Disease; Mixed Dementias; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization allocation to study arms is concealed from all study personnel until the point of randomization assignment.
  In the ADRD-PC Study, the overall PI (Dr. Hanson) and the research staff Clinical Research Coordinators (CRC) collecting data in 30- and 60-day interviews (data source for primary outcome and most secondary outcomes) are masked to study assignment until planned study arm reveal during final analyses. CRCs will conduct 60-day electronic health record (EHR) reviews only after dyads complete study participation, as EHR content has the potential to reveal study arm assignment. As with most behavioral clinical interventions, participants and care providers cannot be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition: ADRD-PC Program (Experimental): 1. Dementia-specific palliative care delivered by hospital-based specialty interdisciplinary palliative care teams.
  2. Standardized caregiver education will be provided by the palliative care team. Clinicians will share and discuss the booklet Advanced Dementia: A Guide for Families, which addresses common concerns and treatment decisions.
  3. Transitional care will be provided by the palliative care team, including facilitation of community-based services and two post-discharge telephone calls.
  Interventions: Behavioral: ADRD-PC Program
- Control Condition (Active Comparator): Patient-family caregiver dyads randomized to the control arm will receive educational materials from the Alzheimer's Association, specifically designed for late-stage ADRD caregivers. The patient will receive usual hospital and post-acute care.
  Interventions: Behavioral: ADRD-PC Program

INTERVENTIONS:
Behavioral: ADRD-PC Program — Included in arm/group descriptions

SUMMARY:
Millions of Americans have late-stage Alzheimer's and related dementias (ADRD), causing suffering due to loss of awareness of self and family, progressive dependency, physical and neuropsychiatric symptoms, and physical, emotional and financial strain for caregivers. Investigators now propose a multi-site randomized clinical trial of the ADRD Palliative Care (ADRD-PC) program for persons with late-stage ADRD and their family caregivers, triggered during hospitalization. Investigators aim to learn if this program of dementia-specific palliative care, standardized caregiver education, and transitional care is effective to reduce burdensome hospital transfers, improve symptom treatment and control, augment supportive services, and reduce nursing home transitions for patients, and to improve caregiver outcomes of communication, shared decision-making and distress.

DETAILED DESCRIPTION:
Investigators have designed the ADRD Palliative Care (ADRD-PC) program of dementia-specific palliative and transitional care, and shown its feasibility and potential efficacy. Delivered by interdisciplinary hospital palliative care teams, ADRD-PC addresses 1) prognostic awareness, 2) symptom management, 3) shared decision-making, and 4) transition to community support services.

The research objective is to conduct a multi-site efficacy randomized clinical trial (RCT) of the ADRD-PC program. Investigators will enroll 424 dyads of hospitalized patients with late-stage ADRD (Global Deterioration Scale (GDS) 6-7 or GDS 5 with significant co-morbidity) with their family caregivers, and an additional 50 dyads that identify as Hispanic/Latino at 5 geographically diverse sites of the Palliative Care Research Cooperative group - University of North Carolina, University of Colorado, Massachusetts General Hospital (Harvard University), Indiana University, and Emory University. The primary hypothesis is that ADRD-PC will reduce hospital transfers (Aim 1). Additional hypotheses are that ADRD-PC will improve patient-centered outcomes of symptom treatment, symptom control, use of community palliative care or hospice, and nursing home transitions (Aim 2); and caregiver outcomes of communication, decision-making and distress (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

People with ADRD Inclusion Criteria:

* aged 55 or older
* hospitalized
* have a physician-confirmed diagnosis of ADRD
* staged GDS 6 or 7; or GDS 5 with additional co-morbidity defined by Charlson Comorbidity Index scored 5 or higher

Caregiver Inclusion Criteria:

* the adult (aged 18 or older) legally authorized representative (LAR) for healthcare and have capacity to serve in this role
* support the person with ADRD
* can complete interviews in English or Spanish.

Exclusion Criteria:

Dyads will be excluded if

* the LAR is not a family caregiver
* the patient currently receives palliative care or hospice
* patient or caregiver would be unduly stressed
* dyad is not successfully randomized.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Hanson, MD, MPH, Principal Investigator — University of North Carolina
Locations (5):
- United States (5):
  - University of Colorado Denver, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. In addition, every attempt will be made to publish results in peer-reviewed journals. Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: 9 to 36 months following publication
Access Criteria: Data may be requested to achieve aims in an approved proposal by contacting the Palliative Care Research Collaborative Group Data Repository.

REFERENCES:
- [Derived] Toles M, Kistler C, Lin FC, Lynch M, Wessell K, Mitchell SL, Hanson LC. Palliative care for persons with late-stage Alzheimer's and related dementias and their caregivers: protocol for a randomized clinical trial. Trials. 2023 Sep 25;24(1):606. doi: 10.1186/s13063-023-07614-4. PMID 37743478

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Condition: ADRD-PC Program: Patient-family caregiver dyads randomized to the intervention arm received ADRD-PC Program during hospitalization and post-acute care.
  1. Dementia-specific palliative care delivered by hospital-based specialty interdisciplinary palliative care teams.
  2. Standardized caregiver education will be provided by the palliative care team. Clinicians will share and discuss the booklet Advanced Dementia: A Guide for Families, which addresses common concerns and treatment decisions.
  3. Transitional care will be provided by the palliative care team, including facilitation of community-based services and two post-discharge telephone calls.
- Control Condition: Patient-family caregiver dyads randomized to the control arm received educational materials from the Alzheimer's Association, specifically designed for late-stage ADRD caregivers. The patients will receive usual hospital and post-acute care.
Period: Overall Study
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Started | 442 | 442
Patients Started | 221 | 221
Caregivers Started | 221 | 221
Completed | 372 | 376
Not Completed | 70 | 66

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition | Total
Number analyzed (Participants) | 442 | 442 | 884
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data are reported separately for Patients and Caregivers.
  years
    Patients: number analyzed (Participants) | 221 | 221 | 442
    Patients | 82.8 (8.03) | 82.5 (7.78) | 82.6 (7.89)
    Caregivers: number analyzed (Participants) | 221 | 221 | 442
    Caregivers | 58.2 (12.9) | 59.5 (12.2) | 58.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are reported separately for Patients and Caregivers.
  Participants
    Patients: number analyzed (Participants) | 221 | 221 | 442
    Patients: Female | 135 | 137 | 272
    Patients: Male | 86 | 84 | 170
    Caregivers: number analyzed (Participants) | 221 | 221 | 442
    Caregivers: Female | 152 | 154 | 306
    Caregivers: Male | 69 | 67 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Patients and Caregivers.
  Participants
    Patients: number analyzed (Participants) | 221 | 221 | 442
    Patients: Hispanic or Latino | 13 | 21 | 34
    Patients: Not Hispanic or Latino | 208 | 200 | 408
    Patients: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 221 | 221 | 442
    Caregivers: Hispanic or Latino | 16 | 18 | 34
    Caregivers: Not Hispanic or Latino | 205 | 203 | 408
    Caregivers: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Patients and Caregivers.
  Participants
    Patients: number analyzed (Participants) | 221 | 221 | 442
    Patients: American Indian or Alaska Native | 0 | 0 | 0
    Patients: Asian | 6 | 2 | 8
    Patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patients: Black or African American | 57 | 55 | 112
    Patients: White | 148 | 146 | 294
    Patients: More than one race | 1 | 4 | 5
    Patients: Unknown or Not Reported | 9 | 14 | 23
    Caregivers: number analyzed (Participants) | 221 | 221 | 442
    Caregivers: American Indian or Alaska Native | 1 | 0 | 1
    Caregivers: Asian | 3 | 3 | 6
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 53 | 57 | 110
    Caregivers: White | 149 | 144 | 293
    Caregivers: More than one race | 2 | 3 | 5
    Caregivers: Unknown or Not Reported | 13 | 14 | 27
Region of Enrollment [Count of Participants; unit: Participants] — Data are reported separately for Patients and Caregivers.
  Participants
    United States: Patients | 221 | 221 | 442
    United States: Caregivers | 221 | 221 | 442

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hospital Transfers (Patients)
Description: Number of hospital transfers (number of emergency room visits + number of hospital admissions )/(person-days of follow-up) within 60 days after discharge from the index hospitalization.
Time Frame: 60 days post index hospital discharge
Measure: Number; unit: events per person day at risk
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
events per person day at risk | 0.99 | 1.12
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.522, Poisson regression

2. Secondary Outcome: Symptom Treatment (Patients)
Description: Palliative Care Domain Index items - 10 items scored present vs absent, scored ranging 0-10 with higher scores indicating increased symptom treatment
Time Frame: 60 days post hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
score on a scale | 8.06 (2.14) | 6.49 (2.27)
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Symptom Control for Physical Symptoms (Patients)
Description: Symptom Management at the End of Life in Dementia (SM-EOLD) - Likert scale, 9 items each scored 0-5, range of 0-45 with higher scores indicating greater symptoms.
Time Frame: 60 days post hospital discharge
Population: Caregivers who skipped questions or did not complete the post hospital discharge follow-up interview are not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 194 | 197
score on a scale | 21.0 (9.08) | 21.8 (9.25)
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.402, t-test, 2 sided

4. Secondary Outcome: Symptom Control for Neuropsychiatric Symptoms-Severity (Patients)
Description: Neuropsychiatric Inventory Questionnaire (NPI-Q) Severity Score - 12 items, each symptom reported as present is rated from 1 (mild) to 3 (severe). The range in this subscale is 0-36 with higher scores indicating worse symptom control.
Time Frame: 60 days post hospital discharge
Population: Caregivers who skipped questions or did not complete the post hospital discharge follow-up interview are not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 192 | 199
score on a scale | 21.6 (5.83) | 21.8 (5.87)
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.803, t-test, 2 sided

5. Secondary Outcome: Symptom Control for Neuropsychiatric Symptoms-Distress (Patients)
Description: Neuropsychiatric Inventory Questionnaire (NPI-Q) Distress - 12 items, if the symptom was reported as present the caregiver rated the level of distress they experienced related tot he patient's symptom from 0 (not distressing) to 5 (extremely distressing). This subscale ranges from 0-60, with higher scores indicating more caregiver distress.
Time Frame: 60 days post hospital discharge
Population: Caregivers who skipped questions or did not complete the post hospital discharge follow-up interview are not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 192 | 199
score on a scale | 24.9 (13.7) | 27.7 (13.8)
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.045, t-test, 2 sided

6. Secondary Outcome: Access to Hospice (Patients)
Description: Percent of people with ADRD who access hospice services.
Time Frame: 60 days post hospital discharge
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
percentage of participants | 17.2 | 17.6
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.977, Chi-squared

7. Secondary Outcome: Access to Community-based Palliative Care (Patients)
Description: Percent of people with ADRD who access community-based palliative care services
Time Frame: 60 days post hospital discharge
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
percentage of participants | 12.7 | 5.9
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.010, Chi-squared

8. Secondary Outcome: Transition to Nursing Home Level of Care (Patients)
Description: Percent of people with ADRD who transition to nursing home care
Time Frame: 60 days post hospital discharge
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
percentage of participants | 35.7 | 36.7
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.935, Chi-squared

9. Secondary Outcome: Documented Discussion of Dementia Prognosis (Patients)
Description: Percent of patients with documented discussion of dementia prognosis in their medical record.
Time Frame: 60 days post hospital discharge
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
percentage of participants | 80.1 | 14.9
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p < 0.001, Chi-squared

10. Secondary Outcome: Documented Discussion of Goals of Care (Patients)
Description: Percent of patients with documented discussion of overall goals of care.
Time Frame: 60 days post hospital discharge
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
percentage of participants | 86.9 | 44.8
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p < 0.001, Chi-squared

11. Secondary Outcome: Shared Decision-making - Hospitalization (Patients)
Description: Percent of patients whose caregivers reported shared decision-making discussions with a healthcare provider about future hospitalization for the patient.
Time Frame: 60 days post hospital discharge
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
percentage of participants | 21.7 | 25.8
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.417, Chi-squared

12. Secondary Outcome: Shared Decision-making - Burdensome Treatment (Patients)
Description: Percent of patients whose caregivers reported shared decision-making about resuscitation, ventilator use, tube feeding, antibiotics for infection treatment.
Time Frame: 60 days post hospital discharge
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 221 | 221
percentage of participants | 38.5 | 42.1
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.531, Chi-squared

13. Secondary Outcome: Caregiver Distress Score (Caregivers)
Description: Family Distress in Advanced Dementia scale - 21 item Likert scale (1=Never to 5=Always) ranges from 21 to 105 with higher scores indicating more distress.
Time Frame: 60 days post hospital discharge
Population: Caregivers who skipped questions or did not complete the post hospital discharge follow-up interview are not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 198 | 200
score on a scale | 48.5 (14.0) | 52.3 (15.4)
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.012, t-test, 2 sided

14. Secondary Outcome: Caregiver Burden (Caregiver)
Description: Zarit Burden scale, short form - 6 items, Likert (1=never to 5=Nearly Always), range 0-24 with higher scores indicating more caregiver burden.
Time Frame: 60 days post hospital discharge
Population: Caregivers who skipped questions or did not complete the post hospital discharge follow-up interview are not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Condition: ADRD-PC Program | Control Condition
Number analyzed (Participants) | 198 | 199
score on a scale | 7.52 (5.44) | 7.44 (5.19)
Statistical Analysis 1: Comparison: Intervention Condition: ADRD-PC Program vs Control Condition; Test type: Superiority; p = 0.876, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from when participants entered the study to 60 days post hospital discharge.
Description: Due to the severity of illness present in the study population, adverse events including mortality and caregiver emotional distress were expected but adjudicated as unrelated to study participation.
Groups:
- Intervention Condition: ADRD-PC Program (Patients): Patients randomized to the intervention arm received ADRD-PC Program during hospitalization and post-acute care.
  1. Dementia-specific palliative care delivered by hospital-based specialty interdisciplinary palliative care teams.
  2. Standardized caregiver education will be provided by the palliative care team. Clinicians will share and discuss the booklet Advanced Dementia: A Guide for Families, which addresses common concerns and treatment decisions.
  3. Transitional care will be provided by the palliative care team, including facilitation of community-based services and two post-discharge telephone calls.
- Intervention Condition: ADRD-PC Program (Caregivers): Caregivers randomized to the intervention arm received ADRD-PC Program during hospitalization and post-acute care.
  1. Dementia-specific palliative care delivered by hospital-based specialty interdisciplinary palliative care teams.
  2. Standardized caregiver education will be provided by the palliative care team. Clinicians will share and discuss the booklet Advanced Dementia: A Guide for Families, which addresses common concerns and treatment decisions.
  3. Transitional care will be provided by the palliative care team, including facilitation of community-based services and two post-discharge telephone calls.
- Control Condition (Patients): Patients randomized to the control arm received educational materials from the Alzheimer's Association, specifically designed for late-stage ADRD caregivers. The patients will receive usual hospital and post-acute care.
- Control Condition (Caregivers): Caregivers randomized to the control arm received educational materials from the Alzheimer's Association, specifically designed for late-stage ADRD caregivers. The patients will receive usual hospital and post-acute care.
Arm/Group | Intervention Condition: ADRD-PC Program (Patients) | Intervention Condition: ADRD-PC Program (Caregivers) | Control Condition (Patients) | Control Condition (Caregivers)
All-Cause Mortality (participants affected / at risk) | 41/221 | 0/221 | 40/221 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/221 | 0/221 | 0/221
Other Adverse Events (participants affected / at risk) | 0/221 | 24/221 | 0/221 | 40/221
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Condition: ADRD-PC Program (Patients) (N=221) | Intervention Condition: ADRD-PC Program (Caregivers) (N=221) | Control Condition (Patients) (N=221) | Control Condition (Caregivers) (N=221)
Emotional Distress (Psychiatric disorders) | 0 (0) | 24 (32) | 0 (0) | 40 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04948866/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT04948866/ICF_000.pdf